CLINICAL TRIAL: NCT00291707
Title: A Phase I Trial of Cetuximab (C225) and Pemetrexed With Concurrent Radiation in Head and Neck Cancer
Brief Title: Trial of Cetuximab and Pemetrexed With Radiation in Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-005
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Head and Neck Cancer
Keywords: head; neck; Cetuximab; Pemetrexed
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Cetuximab; Pemetrexed; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab — The initial dose of cetuximab is 400 mg/m2 intravenously administered over 120 minutes, followed by weekly infusions at 250 mg/m2 IV over 60 minutes. The infusion rate of cetuximab must never exceed 5 mL/min.
  Other Names: C225; ERBITUX
Drug: Pemetrexed — • Pemetrexed 350-500 mg/m2 IV over 10 minutes (see dose escalation design. Dose will be decreased to 200 mg/m2, if the first dose level of 350 mg/m2 is not tolerable) on days 1 and 22, (and 43 if >6000 cGy to be delivered)
  Other Names: ALIMTA
Procedure: radiation therapy — • Radiation therapy standard fractionation 2 Gy/day without planned interruptions beginning on day 1. Radiation will be given M-F for 6-7 consecutives weeks

SUMMARY:
The purpose of this Phase I study is to determine the safety and effectiveness of two chemotherapies drugs, Cetuximab and Pemetrexed (Alimta), when given in combination with radiation therapy.

DETAILED DESCRIPTION:
The purpose of this Phase I study is to determine the safety and effectiveness of two chemotherapies drugs, Cetuximab and Pemetrexed (Alimta), when given in combination with radiation therapy. Currently Pemetrexed is approved by the Food and Drug Administration (FDA) for two other types of cancer, mesothelioma and lung cancer, but it is considered investigational and is not approved by the FDA for head and neck cancer. Cetuximab is approved by the FDA for the treatment of colorectal cancer; however, it is not yet approved for head and neck cancer.

Pemetrexed is a drug that kills tumor cells by stopping cells from functioning normally. It has been studied in thousands of subjects and has been shown to be effective at killing tumor cells in many cancers, including head and neck cancer. In preclinical studies, Pemetrexed showed such promising activity against a wide range of tumor types including those mentioned above as well as breast, colon, and bladder cancers.

Cetuximab (also known as "C225" and "Erbitux") can increase the effectiveness of our standard treatment with chemotherapy and radiation. Cetuximab is a type of drug known as a monoclonal antibody. Monoclonal antibodies are used to try to destroy some types of cancer cells while causing little harm to normal cells. They are designed to recognize specific molecules that are on the surface of particular cancer cells. The monoclonal antibody recognizes the protein and locks onto it. This may trigger the body's immune system to attack the cancer cells and can sometimes make the cells destroy themselves. Cetuximab targets the epidermal growth factor receptor (EGFR), an important molecule for the growth of cancer cells. The use of radiation therapy and Cetuximab has also been studied with good results. We will find what effects (good and bad) Cetuximab has on you and your head and neck cancer.

Both Cetuximab and Pemetrexed have been studied intensively to determine their effectiveness.

In this study, we will find what effects (good and bad) Cetuximab and Pemetrexed, with radiation; have on you and on your head and neck cancer. We will find out if the combination of Cetuximab, Pemetrexed and radiation has better results than what we ordinarily expect with radiation and chemotherapy. We will also find out if the side effects are worse than those we usually see. In addition, we will test both blood and tumor tissue and determine what effects Cetuximab has on these specimens. Finally, we will look for "markers," or cancer identifiers, in your tumor cells and blood that may help to predict what the best treatment is for head and neck cancer patients in the future.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed head and neck malignancy
* All subjects requiring radiotherapy to the head and neck for a poor-prognosis malignancy will be eligible.
* Two cohorts of subjects: no prior history of head and neck radiation, i.e. non-irradiated and prior history of head and neck radiation, i.e. previously irradiated.
* Subjects with recurrent head and neck cancer with no clinically measurable distant disease as well as those subjects in whom distant disease was of low volume and local and regional palliation is clinically warranted will be eligible.
* Subjects without prior treatment should have stage IV disease (see AJCC staging system in Appendix 2, Protocol) or have an expected long-term survival of less than 10%.
* No prior treatment with systemic anti-EGFR inhibitors or Pemetrexed. Any number of prior systemic therapies is allowed.
* Measurable or evaluable disease.
* ECOG performance status 0-2 .
* Age ³ 18 years.
* Subjects must have fully recovered from the effects of any prior surgery, chemotherapy, or radiation therapy. A minimum time period of 4 weeks should elapse between the completion of prior chemotherapy and enrollment in the study.
* ANC ³ 1500/µl, platelet count ³ 100,000/µl. Hemoglobin should be >8 g/dL.
* Creatinine clearance 45 ml/min or higher calculated using the Cockcroft-Gault formula: Calculated Creatinine Clearance = (140-age) X actual body wt.(kg) 72 X serum creatinine Multiply this number by 0.85 if the subject is female
* Total bilirubin within normal limits and AST/ALT less than 3 times the upper limit of normal (less than 5 times the upper limit of normal in the presence of liver metastases).
* Informed consent must be obtained from all subjects prior to beginning therapy. Subjects should have the ability to understand and the willingness to sign a written informed consent document.
* Subjects should be willing and able to take folic acid and vitamin B12 supplementation and should interrupt aspirin or other nonsteroidal anti-inflammatory agents for a 5-day period (8-day period for long acting agents such as piroxicam), see section 5.57

Exclusion criteria:

* Subjects with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would limit compliance with study requirements, significant history of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 3 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* May not be receiving any other investigational agents.
* Pregnant women are excluded from this. Breastfeeding should be discontinued if the mother is treated with chemotherapy. Prior to study enrollment, women of childbearing potential (WOCBP) must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control. Subjects who are women of childbearing potential and sexually active males must be willing to use effective contraception while on study.
* All WOCBP should be instructed to contact the Investigator immediately if they suspect they might be pregnant .
* HIV-positive subjects are excluded from the study.
* Prior grade 3 or 4 infusion or hypersensitivity reaction to a monoclonal antibody.
* For subjects who have baseline clinically significant pleural or peritoneal effusions before initiation of protocol therapy, consideration should be given to draining the effusion prior to starting therapy due the potential of increased toxicity with Pemetrexed in that setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-03; Primary Completion 2008-03 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the maximum tolerated doses and dose-limiting toxicities of Pemetrexed and Cetuximab when given concurrently with radiation in poor prognosis subjects with head and neck cancer. | 10 years

SECONDARY OUTCOMES:
To evaluate the objective response rate post chemoradiotherapy (in subjects with measurable disease), time to progression, and overall survival with the above therapy. | 10 years
To collect tumor tissue from pretreatment biopsies for future biomarker studies and to collect pre- and post-therapy blood samples for future studies, that may include analysis of DNA and RNA extracted from these samples. | indefinite

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Bauman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States